CLINICAL TRIAL: NCT04565886
Title: Clinical and Radiographic Outcomes Following Non-surgical Mechanical Therapy of Peri-implantitis With or Without Adjunctive Diode Laser Application: A 12-month Double-blinded Randomized Clinical Trial
Brief Title: Non-surgical Mechanical Therapy of Peri-implantitis With or Without Adjunctive Diode Laser Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-01163
Record Dates: First submitted 2020-09-22; First posted 2020-09-25 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: Randomised placebo controlled monocentric trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (Sham Comparator): Non-surgical mechanical instrumentation 3x. Each time the laser will be held in place but will not be activated.
  Interventions: Device: Sham Diode laser
- laser (Experimental): Non-surgical mechanical instrumentation 3x with adjunctive diode laser application according to the protocol of the Department of Periodontology, University of Bern
  Interventions: Device: Diode laser application

INTERVENTIONS:
Device: Diode laser application — After mechanical debridement, the pockets around the implant will be rinsed with sterile saline solution. Adjunctive diode laser (settings: 810 nm, 2.5 W, 50 Hz, 10 ms) will be applied 3x for 30 s (i.e., 90 s per appointment) using a 400-lm thick fiber (WhiteStar, Orcos Medical AG, Küsnacht, Switzerland) in the test group. In the control group, non-activated (= placebo) adjunctive diode laser will be applied. The entire treatment procedure, including mechanical debridement, will be performed at Day 0 (= baseline), 7 and 14. The laser decontamination procedure will occur by systematically moving the laser tip along the subgingival implant surface in a vertical and horizontal scanning way. The laser tip will be checked after 4-5 s for coagulation to prevent hotspots in the soft tissues.
  Arms: laser
Device: Sham Diode laser — After mechanical debridement, the pockets around the implant will be rinsed with sterile saline solution. Non-activated (= placebo) adjunctive diode laser will be applied. The entire treatment procedure, including mechanical debridement, will be performed at Day 0 (= baseline), 7 and 14. The laser decontamination procedure will occur by systematically moving the laser tip along the subgingival implant surface in a vertical and horizontal scanning way.
  Arms: control

SUMMARY:
Peri-implantitis is a pathological condition occurring in tissues around dental implants, characterized by inflammation in the peri-implant connective tissue and progressive loss of supporting bone. The goals of peri-implantitis treatment is the resolution of peri-implant soft tissue inflammation and stabilization of the bony attachment (e.g., the level of osseointegration). For this decontamination of the implant surface is mandatory. In order to increase implant surface decontamination, several adjunctive tools have been proposed and investigated both in pre-clinical and clinical studies such as the use of photodynamic therapy and lasers. So far, no data are available to clearly demonstrate the efficacy of the adjunctive use of a diode laser in the non-surgical treatment of peri-implantitis. Therefore, the aim of the present randomized controlled trial (RCT) is to investigate the adjunctive effect of the application of a diode laser to treat peri-implantitis lesions by means of a non-surgical approach. A total of 30 patients is randomly allocated to two groups. The test group receives 3 x nonsurgical mechanical treatment with diode laser application whereas the control group receives the same treatment with sham laser application. The primary outcome is the peri-implant pocket probing depth at 12 months.

DETAILED DESCRIPTION:
Peri-implantitis is a pathological condition occurring in tissues around dental implants, characterized by inflammation in the peri-implant connective tissue and progressive loss of supporting bone. Peri-implantitis is a disease with increasing incidence that, if left untreated, leads to implant loss. The etiological factors of peri-implant infections are similar to those involved in periodontal diseases. Consequently, the goals of peri-implantitis treatment must be the resolution of peri-implant soft tissue inflammation and stabilization of the bony attachment (e.g., the level of osseointegration). This can only be achieved under the condition that the majority of bacterial biofilms and hard deposits are eliminated on the implant surface to create a biologically acceptable surface conducive to wound healing. Decontamination of the implant surface is mandatory to resolve the inflammatory process and to establish healthy peri-implant tissues. To increase implant surface decontamination, several adjunctive tools have been proposed and investigated both in pre-clinical and clinical studies such as the use of photodynamic therapy and lasers. So far, no data are available to clearly demonstrate the efficacy of the adjunctive use of a diode laser in the non-surgical treatment of peri-implantitis. Therefore, the aim of the present randomized controlled trial (RCT) is to investigate the adjunctive effect of the application of a diode laser to treat peri-implantitis lesions by means of a non-surgical approach. A total of 30 patients is randomly allocated to two groups. The test group receives 3 x nonsurgical mechanical treatment with diode laser application whereas the control group receives the same treatment with sham laser application. The primary outcome is the mean peri-implant pocket probing depth (PPD) at 12 months. The secondary endpoints are:

* Change at deepest PPD (mm)
* Change in probing attachment level (PAL) (mm)
* Change in the % of implants with BoP / SUP
* Mean radiographic bone fill (mm) at mesial and distal sites
* Change in width of keratinized mucosa (KM) (mm)
* Change in microbial samples composition at 6 and 12 months
* Changes in patients' related outcomes measures (PROMs) by means of a Visual Analogue Scale (VAS) (range: 0-10)
* Change in peri-implant crevicular fluid (PICF) composition

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy patients enrolled in regular supportive periodontal therapy (SPT)
* Tissue level (TL) implants with an SLA surface supporting single-unit crowns (SUCs) or fixed dental prostheses (FDPs)
* Pocket Probing Depth (PPD) > 5 mm
* Presence of BoP and /or SU
* Radiographic evidence of crestal bone loss ≤ 2mm based on periapical radiographs after delivery of the final restoration
* Cleansable cemented or screw-retained restoration
* Presence of at least 2 mm of keratinized and attached mucosa (KM)
* Signed informed consent

Exclusion Criteria:

* Systemic diseases that could interfere with the treatment outcome (e.g. uncontrolled diabetes mellitus, chemotherapy, etc.)
* Previous peri-implantitis treatment
* Full-Mouth Plaque Score (FMPS) > 25%
* Full-Mouth Bleeding Score (FMBS) > 25%
* Cigarette smoking > 10 cig./day
* Removable implant-supported restorations
* Implant mobility

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Change in peri-implant pocket probing depth (PPD) | at 12 months
  the difference between baseline PPD and PPD after 12 months

SECONDARY OUTCOMES:
Change at deepest PPD (mm) | at 12 months
  Difference of baseline and final PPD of the deepest measurment
Change in probing attachment level (PAL) (mm) | at 12 months
  Difference of attachment level from baseline to 12 months
Change in the % of implants with BoP / SUP | at 12 months
  Difference between baseline and final BoP
Mean radiographic bone fill (mm) at mesial and distal sites | at 12 months
  the distance from the implant shoulder to the bone crest
Change in width of keratinized mucosa (KM) (mm) | at 12 months
  the difference between the baseline and final amount of KM
Change in microbial samples composition | at 6 and 12 months
Changes in patients' related outcomes measures (PROMs) by means of a Visual Analogue Scale (VAS) (range: 0-10) | at 12 months
Change in peri-implant crevicular fluid (PICF) composition | at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Periodontology, University of Bern, Bern, Switzerland